CLINICAL TRIAL: NCT04920721
Title: Retrospective Study of Immediate Hypersensitivity (IHS) Reactions to Platinum Salts in the University Hospital of Nancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, ADAM Tania, Dr, Central Hospital, Nancy, France
Other Study IDs: 2021PI002
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Drug Allergy
Keywords: immediate hypersensitivity; platinum salts; skin tests; tolerance induction
MeSH Terms: conditions — Drug Hypersensitivity; Hypersensitivity, Immediate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Allergic: suspected of immediate hypersensitivity reaction to platinum salts with positiv skin tests
  Interventions: Other: no intervention
- Non allergic: suspected of immediate hypersensitivity reaction to platinum salts with negativ skin tests
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention descriptiv study

SUMMARY:
To assess the efficacy of skin tests with platinum salts in patients suspects with immediate hypersensitivity reactions.

All patients adressed in consultation to the Allergy Department of university hospital of nancy for an immediate hypersensitivity reaction to platinum salts between 2015 and 2021 were retrospectively recruited.

ELIGIBILITY:
Inclusion Criteria:

* adult
* suspected immediate hypersensitivity reaction to platinum salts

Exclusion Criteria:

* skin tests not achievable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with suspected immediate hypersensitivity reactions to platinum salts
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Result of skin test | baseline
  prick test and if negativ => intradermoreaction

CONTACTS AND LOCATIONS:
Overall Officials: Tania ADAM, Dr, Principal Investigator — CHRU Nancy
Locations (1):
- CHRU Nancy, Nancy, Vandoeuvre-Lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No